CLINICAL TRIAL: NCT00863330
Title: A Phase II Study Using Short-Term Cultured Anti-Tumor Autologous Lymphocytes Following a Non-Myeloablative Lymphocyte Depleting Chemotherapy Regimen in Metastatic Melanoma
Brief Title: Laboratory-Treated Autologous Lymphocytes and Aldesleukin After Cyclophosphamide and Fludarabine in Treating Patients With Metastatic Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: administrative decision- PI retired and treating physician left the institution
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000636885; STLMC-L-0839
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Results first posted 2014-12-17 (Estimated); Last update posted 2024-10-03 (Actual); Status verified 2014-12

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Determine toxicity of treatment regimen. (Experimental)
  Interventions: Biological: Tumor Infiltrating Lymphocytes (TIL)

INTERVENTIONS:
Biological: Tumor Infiltrating Lymphocytes (TIL) — Tumor harvest process tumor infiltrating lymphocytes. Non myeloblative chemotherapy consisting of cyclophosphamide and fludarabine. Infusion of TIL cells followed by high dose IL-2.

SUMMARY:
RATIONALE: Treating lymphocytes in the laboratory may help the lymphocytes kill more tumor cells when they are put back in the body. Aldesleukin may stimulate the lymphocytes to kill tumor cells. Drugs used in chemotherapy, such as cyclophosphamide and fludarabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving laboratory-treated lymphocytes and aldesleukin together with cyclophosphamide and fludarabine may kill more tumor cells.

PURPOSE: This phase II trial is studying how well laboratory-treated autologous lymphocytes and aldesleukin work when given after cyclophosphamide and fludarabine in treating patients with metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the ability of treatment with short-term cultured autologous tumor-infiltrating lymphocytes (TIL) in combination with high-dose aldesleukin after a nonmyeloablative lymphocyte-depleting preparative regimen comprising cyclophosphamide and fludarabine phosphate to mediate tumor regression in patients with metastatic melanoma.
* Determine the toxicity of this treatment regimen.

Secondary

* Determine the rate of repopulation of the young TIL cells.
* Establish in vitro immunological correlates that predict in vivo persistence and clinical response.

OUTLINE:

* Conditioning regimen: Patients receive cyclophosphamide IV over 1 hour on days -7 and -6 and fludarabine phosphate IV over 30 minutes on days -5 to -1.
* Tumor-infiltrating lymphocyte (TIL) infusion and high-dose aldesleukin: Patients receive short-term cultured autologous TIL IV over 20-30 minutes on day 0. Patients also receive high-dose aldesleukin IV over 15 minutes every 8 hours on days 0-4.

Patients with stable disease, partial response, or recurrent disease after initial response may receive 1 additional course of treatment (as above) beginning 8 weeks after completion of aldesleukin.

Blood samples are collected at baseline, at 1 week and 1 month after TIL infusion, and then periodically thereafter for research studies. Samples are analyzed for differences in function and phenotype prior to and after TIL infusion. The immunological correlates of treatment are also evaluated using FACS, cytokine release assays, ELISPOT assays, flow cytometry, and PCR. TIL that are cryopreserved at the time of infusion are analyzed to determine cell phenotype and function; correlation of in vitro characteristics of the infused cells with in vivo antitumor activity; and the activity, specificity, and telomere length using flow FISH.

After completion of study treatment, patients are followed at 4-6 weeks, every 3 months for 1 year, every 6 months for 2 years, and then annually for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of metastatic melanoma
* Refractory to standard treatment including high-dose aldesleukin (IL-2), unless previously ineligible for or refused IL-2
* Measurable disease with ≥ 1 lesion that is resectable for tumor-infiltrating lymphocyte generation
* Patients with ≥ 1 brain metastases < 1 cm each, or 1-2 brain metastases > 1 cm are eligible provided they have been treated and stable for ≥ 3 months

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy > 3 months
* ANC > 1,000/mm^3 (without filgrastim support)
* WBC > 3,000/mm^3
* Hemoglobin > 8.0 g/dL
* Platelet count > 100,000/mm^3
* Serum ALT/AST < 3 times upper limit of normal
* Total bilirubin ≤ 2 mg/dL (< 3 mg/dL in patients with Gilbert's syndrome)
* Serum creatinine ≤ 1.6 mg/dL
* LVEF > 45% in patients meeting the following criteria:

  * Clinically significant atrial and/or ventricular arrhythmias, including, but not limited to, atrial fibrillation, ventricular tachycardia, or second- or third-degree heart block
  * At least 60 years of age
* FEV_1 > 60% in patients meeting the following criteria:

  * Prolonged history of cigarette smoking
  * Symptoms of respiratory dysfunction
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 4 months after completion of study treatment
* No HIV or hepatitis B or C positivity
* No form of primary immunodeficiency (e.g., severe combined immunodeficiency disease or AIDS)
* No opportunistic infections
* No active systemic infections
* No history of severe immediate hypersensitivity reaction to any of the agents used in this study
* No coagulation disorders
* No myocardial infarction, cardiac arrhythmias, or positive stress thallium or comparable test
* No history of coronary revascularization or ischemic symptoms
* No obstructive or restrictive pulmonary disease
* No other active major medical illness of the cardiovascular, respiratory, or immune system

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy (alopecia or vitiligo allowed)
* At least 6 weeks since prior ipilimumab

  * Must have normal colonoscopy with normal colonic biopsies
* At least 4 weeks since prior systemic therapy
* Minor surgical procedures within the past 3 weeks allowed provided all toxicities have recovered to ≤ grade 1
* No concurrent systemic steroids
* No other concurrent experimental agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P. Hanson, MD, Principal Investigator — St. Luke's Medical Center; Jonathan S. Treisman, MD, Principal Investigator — St. Luke's Medical Center
Locations (1):
- Aurora St. Luke's Medical Center, Milwaukee, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 14 participants were enrolled. For those, 8 were screen failures and 6 started the study.
Period: Overall Study
Arm/Group | Determine Toxicity of Treatment Regimen.
Started | 6
Completed | 0
Not Completed | 6
Not completed — study terminated early due to administra | 6

BASELINE CHARACTERISTICS:
Arm/Group | Determine Toxicity of Treatment Regimen.
Number analyzed (Participants) | 6
Age, Customized [Number; unit: participants]
  18 or over | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Primary Objective
Description: Determine the ability of autologous cells infused with minimal in vitro culture in conjunction with high dose interleukin -2 (IL-2) following non-myeloablative lymphodepleting preparative regimen to mediate tumor regression in patients with metastatic melanoma.
Time Frame: 4-6 weeks after completion of TIL
Population: Study was terminated for administrative reasons. complete data was not collected and no data analysis was completed
Arm/Group | Determine Toxicity of Treatment Regimen.
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Determine Toxicity of Treatment Regimen.
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
Study was ended early, before substantial data could be collected, due to Investigators retiring/leaving the institution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes